CLINICAL TRIAL: NCT01698021
Title: Quantification and Description of the Increase in Serum Troponin Following Acute Coronary Syndrome
Acronym: QUANTUM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Other Study IDs: Projet 12-081
Record Dates: First submitted 2012-09-28; First posted 2012-10-02 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2012-09

CONDITIONS: Acute Coronary Syndrome; Myocardial Infarction; Unstable Angina
Keywords: Creatine Kinase, MB form; Troponin; Acute coronary syndrome; myocardial infarction; Unstable angina
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction; Angina, Unstable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The new assay of troponins T (highly sensitive troponins) detects concentrations much lower than before. Few data are currently available on their kinetics during acute coronary syndrome, especially in regard to the correlation with CK MB. The aim of the present study is to describe the kinetic of highly sensitive troponins in acute coronary syndrome, to correlate it with the concentration of CK MB, and possibly to evaluate their prognostic value with respect to infarct size .

DETAILED DESCRIPTION:
Patients who meet the inclusion criteria will have a highly sensitive troponins and CKMB assays q 8hr for the first day, and q 12h for the next 2 days. If clinically not indicated, the blood sample can be cancelled at any time, as in the case of a patient with an initial suspicion of acute coronary syndrome in which the final diagnosis is something else. Only patients with a definitive myocardial infarction will be analyzed.

Subgroup analyses includes ST-elevation MI, Non ST-elevation MI, revascularization vs no revascularization, procedural myocardial infarction.

Another analysis conducted is the correlation between the values of troponin and infarct size by echocardiography (in patients who have an echocardiography 2-7 days post AND 2-6 months post myocardial infarction)

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years-old
* Clinical suspicion of an acute coronary syndrome; (will be analyzed only patients with aposteriori definitive diagnosis of unstable angina or myocardial infarction)

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients presenting to the emergency department or being hospitalized for any reason in which we suspect an acute coronary syndrome.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2013-06; Primary Completion 2013-11 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Evaluation of troponins kinetic in acute coronary syndromes. | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Paul Farand, Md MSc, Principal Investigator — Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Locations (1):
- Centre Hospitalier Universitaire de Sherbrooke, departement de cardiologie, Sherbrooke, Quebec, Canada